CLINICAL TRIAL: NCT01624194
Title: Double-blind, Randomized, Placebo Controlled Trial of Intranasal Oxytocin Treatment for Social Deficits in Children With Autism.
Brief Title: Intranasal Oxytocin Treatment for Social Deficits in Children With Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Antonio Hardan, Associate Professor of Child Psychiatry, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU-12132011-8827
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin nasal spray (Active Comparator): Prior to randomization, all subjects will participate in a 1-week open-label placebo lead-in trial. Each subject will be administered the placebo nasal spray at Stanford University and then their parent will continue administering the nasal spray to the subject for 1 week at home. Each subject will then be randomly assigned either to the active group or to the placebo (stratified by gender) and will be given the appropriate nasal spray bottle and their parents will be responsible for administering 3 puffs per nostril (4 IU/puff) to their child for a total dose of 24 IU oxytocin or placebo twice daily (BID; morning and evening) for 4-weeks. On completion of this 4-week treatment trial subjects will have the option of participating in a second double-blind trial in which they will be assigned to the alternate nasal spray, to that which they received during the first 4-week trial, for an additional 4-week period.
  Interventions: Drug: Oxytocin nasal spray
- Placebo nasal spray (Placebo Comparator): The placebo nasal spray bottles will be prepared by adding all of the ingredients used in the Syntocinon nasal sprays with the exception of the concentrated oxytocin solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin nasal spray — 24IU BID (3 x 0.1 mL [4IU] sprays per nostril twice daily for 4-weeks.
  Other Names: Syntocinon® Nasal Spray
  Arms: Oxytocin nasal spray
Drug: Placebo — 3 x 0.1 mL sprays per nostril twice daily for 4-weeks.
  Arms: Placebo nasal spray

SUMMARY:
Autism is a pervasive developmental disorder characterized by core deficits in social behavior and communication, and the presence of repetitive or stereotyped behaviors. It is one of three recognized disorders in the autism spectrum which affects an estimated 1 in 88 children in the United States. At present, pharmacotherapies target only associated features of autism, with no effective drug treatments for the social impairments. Several lines of evidence now suggest that the neuropeptide oxytocin (OT) may be an effective treatment for the core social deficits in autism. Here we will test the effects of twice daily intranasal OT (24 IU) over a 4-week period for enhancing social deficits in male and female children aged 6-12 years with autism. This research has high potential to lead to the development of more effective treatments and earlier interventions for children with autism.

DETAILED DESCRIPTION:
In recent years, the neuropeptide oxytocin (OT) has been implicated in a wide range of social behaviors including attachment bonds, emotion recognition, eye gaze to social cues, and memory for social information. Social impairments represent one of the most intractable features of autism, and evidence now suggests that OT biology is dysregulated in individuals with this disorder. The central aim of the research outlined here is to test whether OT administration to children with autism increases their quality and quantity of social interactions and enhances their ability to process emotional and social information. Findings from initial single-dose OT administration studies in teenaged and adult males with autism have shown improvement in some aspects of social functioning, but replication and extension to well-controlled treatment trials with younger male and female subjects is necessary to evaluate effectiveness. We therefore aim to investigate the effect of intranasal OT on social cognition and behavior immediately following a single-dose (24IU) and following a 4-week period of OT (24IU BID) administration in a sample of 50 subjects with autism aged 6 to 12 years. The primary outcome for this study is change in social behavior, as determined by parent ratings on the Social Responsiveness Scale (SRS) after the 4-week treatment period. Secondary outcomes are changes in functioning on laboratory-based measures of social behavior and cognition following single-dose and 4-week OT administration. Research in a small study sample (N=13) also identified treatment responders and non-responders to a single-dose of OT. Thus, we also aim to identify biological and cognitive and behavioral variables (i.e., pretreatment levels of social functioning and pretreatment plasma hormone levels) that may influence treatment response efficacy in our larger study sample. On completion of the 4-week treatment period all subjects will have the option of participating in another 4-week double-blind trial in which they will be switched to the alternate nasal spray to that which they previously received. They will then undergo a fourth and final assessment time-point using the same testing procedures as outlined above on completion of the 4-week dosing. By providing subjects with the option of participating in a second 4-week treatment trial, all subjects will have an opportunity to receive the active oxytocin nasal spray. We also will be able to examine any ongoing effects of oxytocin treatment in the group receiving placebo during the second 4-week administration period. Subjects not willing to take part in the second trial will exit the study and will be referred to their treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy outpatients between 6 and 12 years of age (cut off 12 years and 11 months)
* Intelligence Quotient > 40
* Diagnosis of autism spectrum disorder based on the Autism Diagnostic Interview - Revised, Autism Diagnostic Observation Schedule, and DSM-IV criteria
* Clinical Global Impression severity rating of 4 or higher
* Care provider who can reliably bring subject to clinic visits, provide trustworthy ratings, and interacts with the subject on a regular basis
* Stable medications for at least 4 weeks
* No planned changes in psychosocial interventions during the trial
* Willingness to provide blood samples.

Exclusion Criteria:

* Diagnostics and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) diagnosis of schizophrenia, schizoaffective disorder, or psychotic disorder
* Regular nasal obstruction or nosebleeds
* Active medical problems: unstable seizures, significant physical illness (e.g., serious liver, renal, or cardiac pathology)
* Sensitivity to preservatives (in particular E 216, E 218, and chlorobutanol hemihydrate)
* A genetic abnormality (e.g., Fragile X Syndrome)
* Significant hearing or vision impairments
* Habitually drinks large volumes of water
* Pregnancy, breastfeeding, or child birth within the last 6 months
* Sexually active females not using a reliable method of contraception.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Y Hardan, MD, Principal Investigator — Stanford University; Karen J Parker, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Parker KJ, Oztan O, Libove RA, Sumiyoshi RD, Jackson LP, Karhson DS, Summers JE, Hinman KE, Motonaga KS, Phillips JM, Carson DS, Garner JP, Hardan AY. Intranasal oxytocin treatment for social deficits and biomarkers of response in children with autism. Proc Natl Acad Sci U S A. 2017 Jul 25;114(30):8119-8124. doi: 10.1073/pnas.1705521114. Epub 2017 Jul 10. PMID 28696286
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in the Autism and Developmental Disabilities Clinic in the Division of Child and Adolescent Psychiatry at Stanford University. Recruitment began in June 2012 and ended in April 2016.
  Participants were recruited through the Stanford Autism Research Registry, flyers posted in the community, posted online and special events.
Pre-assignment Details: 54 subjects were consented and assessed for eligibility. 19 subjects were excluded (13 did not meet inclusion criteria and 6 declined to participate). Additionally, 1 subject allocated to oxytocin did not receive allocated intervention due to parent declining to participate.
Groups:
- Oxytocin Nasal Spray: Oxytocin nasal spray: 24IU twice daily (BID) (3 x 0.1 mL [4IU] sprays per nostril twice for 4-weeks.
Period: Overall Study
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Started | 16 | 18
Completed | 14 | 18
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Oxytocin Nasal Spray: Oxytocin nasal spray: 24IU BID (3 x 0.1 mL [4IU] sprays per nostril twice for 4-weeks.
- Total: Total of all reporting groups
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 18 | 34
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 14 | 14 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6 | 8 | 14
  Asian | 4 | 5 | 9
  Other | 6 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Parent Rated Social Responsiveness Scale (SRS) Scores During Treatment.
Description: Social Responsiveness Scale (SRS) raw scores measure social abilities with lower raw scores meaning better social abilities. (Raw Score Range: 0 - 195)
Time Frame: Baseline; Week 4
Population: Participants who completed the protocol are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 14 | 18
units on a scale | 9.73 (2.64) | 3.18 (2.18)
Statistical Analysis 1: Comparison: Oxytocin Nasal Spray vs Placebo Nasal Spray; Test type: Other; p = 0.0275, General Linear Model (GLM)

2. Secondary Outcome: Number of Participants With Side Effects Assessed Using Parent Rated Dosage Record Treatment Emergent Symptom Scale (DOTES) Scores During Treatment
Description: Dosage Record Treatment Emergent Symptom Scale (DOTES) side effects reported by parents during 4-weeks of treatment. Participant Counts are used.
Time Frame: Baseline through Week 4
Measure: Number; unit: participants
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 14 | 18
participants
  Cold Symptoms | 0 | 1
  Fever | 0 | 1
  Cough | 1 | 0
  Headache | 1 | 0
  Insomnia | 1 | 1
  Excitement/Agitation | 1 | 2
  Depressive Affect | 0 | 1
  Labile Mood | 1 | 1
  Silly Behavior | 1 | 0
  More Distractible | 1 | 0
  Nasal Congestion | 3 | 0
  Epistaxis | 1 | 0
  Sneezing | 0 | 1
  Mouth Pain | 0 | 1
  Intranasal Swelling | 1 | 0
  Runny Nose | 1 | 0
  Blinking Eyes | 0 | 1
  Earache | 0 | 1
  Nasal Discomfort | 0 | 1
  Loose Stool | 1 | 0
  Constipation | 1 | 0
  Stomach Discomfort | 0 | 1
  Skin Cut | 0 | 2
Statistical Analysis 1: Comparison: Oxytocin Nasal Spray vs Placebo Nasal Spray; Test type: Other; p > 0.05, Fisher Exact — Fisher's Exact Test was used to test for differences in adverse events between oxytocin-treated and placebo-treated individuals. A p-value of ≤0.05 would have been statistically significant

3. Secondary Outcome: Change From Baseline in Height.
Time Frame: Baseline; Week 4
Population: Participants with available data are included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: cm
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 14 | 17
cm
  Baseline | 134 [126 to 141] | 129 [122 to 135]
  Week 4 | 134 [127 to 142] | 129 [122 to 136]
Statistical Analysis 1: Comparison: Oxytocin Nasal Spray vs Placebo Nasal Spray; Test type: Other; p > 0.05, Mixed Models Analysis; A mixed-models analysis was used to compare between groups, and between baseline and Week 4

4. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Score at Week 4
Description: This outcome is reported as the count of participants in each CGI-I rating category at the week 4 visit, assessing change over the 4-week period. CGI-I rating of 1=Very Much Improved, 2=Much Improved, 3=Minimally Improved, 4=No Change, 5=Minimally Worse, 6=Much Worse, and 7=Very Much Worse.
Time Frame: Baseline to Week 4
Population: Participants with available data are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 14 | 18
Participants
  Very Much Improved | 0 | 0
  Much Improved | 3 | 3
  Minimally Improved | 2 | 5
  No Change | 9 | 10
  Minimally Worse | 0 | 0
  Much Worse | 0 | 0
  Very Much Worse | 0 | 0

5. Secondary Outcome: Parent Rated Aberrant Behavior Checklist (ABC) Irritability Scores at Baseline and Week 4
Description: Higher scores indicate more symptoms, lower scores indicate fewer symptoms. Irritability scores can range from 0-45. Lethargy scores can range from 0-48. Stereotypy scores can range from 0-21. Hyperactivity scores can range from 0-48. Inappropriate speech scores can from 0-12.
Time Frame: Baseline; Week 4
Population: Participants with available data are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 16 | 18
units on a scale
  Baseline Irritablity | 13.20 (11.91) | 13.94 (8.71)
  Week 4 Irritability | 8.86 (8.87) | 11.78 (8.11)
  Baseline Lethargy | 14.13 (8.70) | 11.7 (8.34)
  Week 4 Lethargy | 10.6 (4.07) | 7.33 (6.30)
  Baseline Stereotypy | 5.69 (6.20) | 5.61 (4.55)
  Week 4 Stereotypy | 4.86 (5.07) | 5.50 (4.85)
  Baseline Hyperactivity | 15.00 (13.74) | 23.28 (10.74)
  Week 4 Hyperactivity | 10.50 (10.17) | 19.11 (9.68)
  Baseline Inappropriate Speech | 3.94 (3.28) | 5.44 (3.99)
  Week 4 Inappropriate Speech | 2.86 (3.23) | 4.17 (3.31)

6. Secondary Outcome: Change From Baseline in Parent Rated Spence Children's Anxiety Scale (SCAS) During Treatment.
Description: Scale measuring severity of anxiety symptoms. Higher scores mean higher levels of anxiety, lower scores mean lower levels of anxiety. (Raw Score Range: 0 - 114)
Time Frame: Baseline; Week 4
Population: Participants who completed the protocol are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 14 | 18
units on a scale | 1.66 (3.05) | 4.53 (2.21)
Statistical Analysis 1: Comparison: Oxytocin Nasal Spray vs Placebo Nasal Spray; Test type: Other; p = 0.3395, General Linear Model (GLM)

7. Secondary Outcome: Change From Baseline in Vineland Adaptive Behavior Scales, Second Edition - Social and Communication Subscales During Treatment.
Description: Higher Social Standard Score means better social skills, lower Social Standard Score means worse social skills. Higher Communication Standard Score means better communication skills, lower Communication Standard Score means worse communication skills. Standard Scores can range from 20 to 160.
Time Frame: Baseline; Week 4
Population: Participants with available data are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 9 | 12
units on a scale
  Baseline Social Standard Score | 61.4 (12.82) | 67.75 (12.45)
  Week 4 Social Standard Score | 66.11 (16.03) | 70.92 (14.23)
  Baseline Communication Standard Scores | 66.91 (19.60) | 71.80 (17.85)
  Week 4 Communication Standard Scores | 71.33 (11.43) | 78.29 (19.12)

8. Secondary Outcome: Change From Baseline in Laboratory Based Facial Emotion Recognition Abilities During Treatment.
Time Frame: Up to 4 weeks
Population: Data were not collected for this outcome.
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in Laboratory Based Eye-gaze to Social Cues During Treatment.
Time Frame: Baseline; Week 4
Population: Data not collected.
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Reading the Mind in the Eyes Test, Child Version (RMET-child) Scores During Treatment.
Time Frame: Up to 4 weeks
Population: Data were not not collected for this outcome.
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in Laboratory Based Social Mimicry Abilities During Treatment.
Time Frame: Up to 4 weeks
Population: Data were not not collected for this outcome.
Groups:
- Oxytocin Nasal Spray: Oxytocin nasal spray: 24IU BID (3 x 0.1 mL [4IU] sprays per nostril twice
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline in Developmental NEuroPSYchological Assessment (NEPSY-II) Affect Recognition Scores During Treatment.
Description: Higher Affect Recognition scores mean better affect recognition abilities, lower Affect Recognition scores mean worse affect recognition abilities.
  Scores can range from 1 to 19.
Time Frame: Baseline; Week 4
Population: Participants with available data were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 4 | 7
units on a scale
  Baseline Affect Recognition Score | 10 (1.89) | 9.43 (3.78)
  Week 4 Affect Recognition Score | 8.75 (1.5) | 6.43 (4.08)

13. Secondary Outcome: Change From Baseline in Plasma Oxytocin Levels During Treatment.
Description: This outcome originally specified that oxytocin, vasopressin, and cortisol levels would be assessed; however, data on vasopressin and cortisol levels were not collected during the study.
  There are no clinical laboratory tests that establish a normative range for oxytocin. Measurements prior to and following treatment were intended to evaluate oxytocin level as a predictor of response.
Time Frame: Up to 4 weeks
Population: Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 11 | 15
pg/mL
  Baseline | 8.82 (4.67) | 8.66 (3.85)
  Week 4 | 10.36 (3.57) | 8.40 (3.57)

14. Secondary Outcome: Change From Baseline in Parent Rated Repetitive Behavior Scale- Revised (RBS-R) Scores During Treatment.
Description: Higher scores on the Repetitive Behavior Scale- Revised mean higher levels of repetitive and restricted behaviors. (Raw Score Total Range: 0 - 129)
Time Frame: Baseline; Week 4
Population: Only analyzed after 4 weeks.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 14 | 18
units on a scale | 5.68 (3.32) | 5.79 (2.78)
Statistical Analysis 1: Comparison: Oxytocin Nasal Spray vs Placebo Nasal Spray; Test type: Other; p = 0.9757, General Linear Model (GLM)

15. Secondary Outcome: Change From Baseline in Weight
Time Frame: Baseline; Week 4
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 14 | 17
kilograms
  Baseline | 32.7 [27.0 to 39.5] | 28.0 [23.5 to 33.2]
  Week 4 | 33.5 [27.7 to 40.4] | 28.4 [23.9 to 33.7]
Statistical Analysis 1: Comparison: Oxytocin Nasal Spray vs Placebo Nasal Spray; Test type: Other; p > 0.05, Mixed Models Analysis; A mixed-models analysis was used to compare between groups, and between baseline and Week 4

16. Secondary Outcome: Change From Baseline in Heart Rate
Time Frame: Baseline; Week 4
Population: Participants with available data are included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 13 | 14
beats per minute
  Baseline Sitting Heart Rate | 92.5 [83.0 to 101.9] | 92.7 [83.6 to 101.8]
  Post 4 -Week Sitting Heart Rate | 97.1 [87.7 to 106.5] | 101.6 [92.5 to 110.6]
Statistical Analysis 1: Comparison: Oxytocin Nasal Spray vs Placebo Nasal Spray; Test type: Other; p > 0.05, Mixed Models Analysis

17. Secondary Outcome: Change From Baseline in Blood Pressure
Time Frame: Baseline; Week 4
Population: Participants with available data are included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 13 | 14
mmHg
  Baseline Systolic Blood Pressure, Sitting | 104.2 [98.7 to 109.8] | 101.0 [95.6 to 106.4]
  Post 4 -Week Systolic Blood Pressure, Sitting | 111.1 [105.5 to 116.6] | 110.9 [105.6 to 116.3]
  Baseline Diastolic Blood Pressure, Sitting | 64.3 [59.0 to 69.6] | 64.6 [59.4 to 69.7]
  Post 4 -Week Diastolic Blood Pressure, Sitting | 71.4 [66.1 to 76.7] | 68.9 [63.8 to 74.1]
  Baseline Systolic Blood Pressure, Standing | 101.6 [95.2 to 108.1] | 107.7 [101.5 to 113.9]
  Post 4 -Week Systolic Blood Pressure, Standing | 111.6 [105.2 to 118.1] | 105.6 [99.4 to 111.9]
  Baseline Diastolic Blood Pressure, Standing | 63.3 [58.0 to 68.6] | 68.2 [63.1 to 73.3]
  Post 4 -Week Diastolic Blood Pressure, Standing | 70.9 [65.6 to 76.2] | 69.8 [64.7 to 74.9]
Statistical Analysis 1: Comparison: Oxytocin Nasal Spray vs Placebo Nasal Spray; Test type: Other; p > 0.05, Mixed Models Analysis — For all blood pressure analyses

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Oxytocin Nasal Spray | Placebo Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/18
Other Adverse Events (participants affected / at risk) | 11/14 | 12/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxytocin Nasal Spray (N=14) | Placebo Nasal Spray (N=18)
Cold Symptoms (General disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Cough (General disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Excitement/Agitation (Psychiatric disorders) | 1 | 2
Depressive Affect (Psychiatric disorders) | 0 | 1
Labile Mood (Psychiatric disorders) | 1 | 1
Silly Behavior (Psychiatric disorders) | 1 | 0
More Distractible (Psychiatric disorders) | 1 | 0
Nasal Congestion (General disorders) | 3 | 0
Epistaxis (General disorders) | 1 | 0
Sneezing (General disorders) | 0 | 1
Mouth Pain (General disorders) | 0 | 1
Intranasal Swelling (General disorders) | 1 | 0
Runny Nose (General disorders) | 1 | 0
Blinking Eyes (Eye disorders) | 0 | 1
Earache (Ear and labyrinth disorders) | 0 | 1
Nasal Discomfort (General disorders) | 0 | 1
Loose Stool (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Stomach Discomfort (Gastrointestinal disorders) | 0 | 1
Skin Cut (Skin and subcutaneous tissue disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
The final sample was 84% male and was not powered to detect sex differences in treatment response. Participants were permitted to take other medications during the intervention. Many of our outcome measures relied on parent report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No